CLINICAL TRIAL: NCT04793802
Title: Impact of Physiotherapy Session With or Without Non Invasive Ventilation in the Patient Benefiting From High Nasal Flow Oxygenation After Cardiac Surgery: a Pilot Study
Brief Title: Impact of Physiotherapy Session in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, PAYSANT Jean, Clinical Professor, Medical Doctor, Philosophiae Doctor, Central Hospital, Nancy, France
Other Study IDs: 2020PI208
Record Dates: First submitted 2020-12-04; First posted 2021-03-11 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Physical Therapy in Cardiac Surgery Patients
Keywords: Physiotherapy; Cardiac surgery; Lung ultrasound score; Noninvasive ventilation; High flow oxygenation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients benefiting from HIGH-FLOW OXYGENATION + NONINVASIVE VENTILATION: Patients benefiting from high-flow oxygenation will have their physiotherapy session with non-invasive ventilation.
  Interventions: Other: PHYSIO
- Patients benefiting from HIGH-FLOW OXYGENATION: Patients benefiting from high-flow oxygenation will have their physiotherapy session without non-invasive ventilation.
  Interventions: Other: PHYSIO

INTERVENTIONS:
Other: PHYSIO — session of physiotherapy

SUMMARY:
This work consists, first of all, in making an inventory of the physiotherapy of the patient undergoing cardiac surgery under high flow oxygenation at the CHRU NANCY.

Then, in a second step, the impact of the physiotherapy on the lung ultrasound score associated or not with the NIV of the patient under OHD after cardiac surgery will be studied.

The objective is therefore to answer the following research question: what is the impact of a physiotherapy session with or without non-invasive ventilation in patients receiving high flow oxygenation after cardiac surgery on the lung ultrasound score measured by ultrasound?

Main hypothesis: Physiotherapy is associated with NIV when it is prescribed in patients undergoing high flow oxygenation after cardiac surgery.

Secondary hypothesis: Physiotherapy + NIV further improves pulmonary aeration versus physiotherapy + high flow oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Person who has received full information on the organization of the research and has not objected to the use of the data.
* Person benefiting from cardiac surgery programmed on Cardiothoracic Bypass
* Patient under high flow oxygenation
* Age ≥ 18 years old
* 18.5 ≤ BMI ≤ 35 kg/m2
* Conscious and oriented patients: Glasgow 15

Exclusion Criteria:

* Surgical emergencies: grafting, dissections...
* Lumbar drainage in progress
* Beating heart surgery
* Refusal to participate in the study
* Persons referred to in Articles L.1121-8 and L.1122-1-2 of the Public Health Code (minors, person under guardianship, under curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects of the study will be patients who stayed in the Cardiovascular Surgery and Cardiac Transplant Intensive Care Unit at NANCY CHRU from September 15, 2020 to March 15, 2021
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Lung ultrasound score | The time of the event (the 2 measurements + the physiotherapy session) is estimated at 45 minutes.
  Reliable and verified score, subject to international recommendations allowing the physiotherapist to deepen his diagnosis and evaluate the effectiveness of his techniques. Measured on 12 thoracic regions The score (N B1 B2 C) will therefore be calculated according to the level obtained in each zone to determine a score out of 36. The higher the score, the more the lung has a deficit of ventilation.
  A decrease in the objective lung ultrasound score will result in better lung aeration.
  Two lung ultrasound score measurements are realized on one patient. The first measurement is taken on the day of inclusion of the patient in the study at the time of the physiotherapist's assessment before the CPT session. (CPT = Chest Physiotherapy Treatment) The second and last measurement is taken after the CPT session (with or without NIV, depending on the medical prescription).

CONTACTS AND LOCATIONS:
Overall Officials: Jean PAYSANT, MD PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU nancy, Nancy, France